CLINICAL TRIAL: NCT07225348
Title: Treatment of Perioral Wrinkles Using Topical Poly-L-lactic Acid and Microneedling Device
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Skincare Physicians of Chestnut Hill (Other)
Collaborators: Galderma R&D (Industry)
Responsible Party: Principal Investigator, Jessica Labadie, Principal Investigator, Skincare Physicians of Chestnut Hill
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SkincarePCH
Record Dates: First submitted 2025-11-03; First posted 2025-11-06 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Perioral Wrinkles
Keywords: perioral wrinkles; microneedling; poly-L-lactic acid
MeSH Terms: interventions — poly(lactide); New-Fill; Percutaneous Collagen Induction

STUDY DESIGN:
Intervention Model Description: The results of Part I will directly affect Part II:
  * If no PLLA is seen in any of the samples from Part I, then we will NOT proceed to the clinical trial in Part II.
  * If PLLA particles are seen in samples from BOTH protocols, then the clinical trial from part II will proceed as written below.
  * If PLLA particles are only seen in the samples where the PLLA serum was applied FIRST, then we will DROP Arm B in Part II.
  * If PLLA particles are only seen in the samples where the PLLA serum was applied second, then we will DROP Arm A in Part II.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Arm A (Experimental): Topical PLLA applied to perioral region first and then a microneedling treatment performed.
  Interventions: Drug: Poly-L-Lactic Acid; Device: Microneedling
- Arm B (Experimental): A microneedling treatment is first performed and then topical PLLA is applied.
  Interventions: Drug: Poly-L-Lactic Acid; Device: Microneedling

INTERVENTIONS:
Drug: Poly-L-Lactic Acid — Topical PLLA diluted with 8cc of sterile water
  Other Names: Sculptra
Device: Microneedling — Microneedling treatment of the perioral region
  Other Names: Eclipse Skin Pen with glide OR MD needle Pen

SUMMARY:
The first goal of this clinical trial is to learn if topical application of PLLA in conjunction with a microneedling treatment works to treat perioral wrinkles in adults. The second goal is to see whether the application of topical PLLA is more effective before or after a microneedling treatment. The main questions it aims to answer are:

* Is PLLA present within the MN channels from in vivo biopsy samples?
* Is it safe to combine topical PLLA and MN in the treatment of perioral wrinkles, as determined by the incidence and severity of adverse events in healthy subjects?
* Does overall aesthetic and skin texture improve in combining microneedling with topical PLLA in the treatment of mild to moderate perioral wrinkles?
* Is it the treatment of topical PLLA more effective when applied before or after a microneedling treatment.

Researchers will compare the application of PLLA before a microneedling treatment to a microneedling treatment with PLLA application after to see which treatment method is more effective.

Participants will:

- receive 2 treatments spaced 4-6 weeks apart of topical PLLA and microneedling

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant, non-lactating females 40-70 years of age
* Fitzpatrick Skin Type I-IV
* Wrinkle severity graded by the investigator (1-3 on Lemperle scale)
* Able to provide written informed consent, understand and be willing to comply with all study related procedures and follow-up visits
* Signed informed consent obtained before any study-specific procedure is performed.

Exclusion Criteria:

* Lesions suspicious for any malignancy, actinic keratosis, melasma, vitiligo, cutaneous papules/nodules or active inflammatory lesions in the area to be treated
* Tenderness in the treatment rea
* History of keloid formation or hypertrophic scarring
* History of trauma or surgery to the treatment area
* Scar present in the areas to be treated
* Silicone or synthetic material injections in the areas to be treated
* Injection of fat, collagen, hyaluronic acid or other dermal fillers in the areas to be treated within the previous 12 months
* History of treatment with dermabrasion or laser in the areas to be treated within the previous 12 months
* History of treatment with botulinum toxin injections in the areas to be treated within the prior 6 months
* Active smokers (0.5 pack/day) or having quit within 3 months prior treatment
* Active, chronic, or recurrent infection
* History of compromised immune system or currently being treated with immunosuppressive agents
* History of sensitivity to analgesic agents, Aquaphor, topical or local anesthetics
* Excessive sun exposure and use of tanning beds or tanning creams within 30 days prior to treatment
* Treatment with fish oil within 14 days prior to treatment
* Treatment with aspirin or other blood thinning agents within 14 days prior to treatment
* History or presence of any clinically significant bleeding disorder
* Co-morbid condition that in the Investigator's opinion could limit ability to participate in the study or to comply with follow-up requirements
* History of drug and/or alcohol abuse
* Any issue that, at the discretion of the investigator, would interfere with assessment of safety or efficacy or compromise the subject's ability to safely undergo study procedures or give informed consent
* Treatment with an investigational device or agent within 30 days before treatment or during the study period

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Global Aesthetic Improvement Scale (GAIS) | 120 days
  blinded in person GAIS scores

SECONDARY OUTCOMES:
Lemperle Wrinkle Scale | 120 days
  three blinded raters, who will judge scores of pre- and post-treatment photographs using the Lemperle Wrinkle Scale
Lemperle Wrinkle Scale | 120 days
  treating investigator reported score using the Lemperle Wrinkle Scale
Canfield VISIA measurements | 120 days
  wrinkle severity scores as calculated by the computerized Canfield VISIA measurements
GAIS | 120 days
  subject and treating investigator reported score using the GAIS

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 120 days
  the incidence and severity of systemic and cutaneous adverse events
Histologic endpoint | 120 days
  PLLA particles visualized within MN channels on H&E with polariscopic examination
Molecular Endpoint | 120 days
  Molecular testing (Gene Markers)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica G Labadie, MD, Principal Investigator — SkinCare Physicians
Locations (1):
- SkinCare Physicians, Chestnut Hill, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cervantes J, Chang YF, Dover JS, Hernandez Alvarez A, Chung HJ. Laser-Assisted and Device-Assisted Filler Delivery: A Histologic Evaluation. Dermatol Surg. 2023 Sep 1;49(9):865-870. doi: 10.1097/DSS.0000000000003870. Epub 2023 Jun 23. PMID 37389474
- [Background] Tian T, Luo Y, Jiang T, Dong Y, Yu A, Chen H, Gao X, Li Y. Clinical effect of ablative fractional laser-assisted topical anesthesia on human skin: A randomized pilot study. J Cosmet Laser Ther. 2016 Nov;18(7):409-412. doi: 10.1080/14764172.2016.1197404. Epub 2016 Aug 5. PMID 27419471
- [Background] Taudorf EH. Laser-assisted delivery of topical methotrexate - in vitro investigations. Dan Med J. 2016 Jun;63(6):B5254. PMID 27264947
- [Background] Waibel JS, Wulkan AJ, Shumaker PR. Treatment of hypertrophic scars using laser and laser assisted corticosteroid delivery. Lasers Surg Med. 2013 Mar;45(3):135-40. doi: 10.1002/lsm.22120. Epub 2013 Mar 4. PMID 23460557
- [Background] Ibrahim O, Ionta S, Depina J, Petrell K, Arndt KA, Dover JS. Safety of Laser-Assisted Delivery of Topical Poly-L-Lactic Acid in the Treatment of Upper Lip Rhytides: A Prospective, Rater-Blinded Study. Dermatol Surg. 2019 Jul;45(7):968-974. doi: 10.1097/DSS.0000000000001743. PMID 30608292
- [Background] Rkein A, Ozog D, Waibel JS. Treatment of atrophic scars with fractionated CO2 laser facilitating delivery of topically applied poly-L-lactic acid. Dermatol Surg. 2014 Jun;40(6):624-31. doi: 10.1111/dsu.0000000000000010. PMID 24852466
- [Background] Physicochemical Characteristics and Hydrolytic Degradation of Polylactic Acid Dermal Fillers: A Comparative Study Nikita G. Sedush 1,* , Kirill T. Kalinin 1, Pavel N. Azarkevich 1 and Antonina A. Gorskaya
- [Background] Courderot-Masuyer C, Robin S, Tauzin H, et al. Evaluation of the behaviour of wrinkles fibroblasts and normal aged fibroblasts in the presence of poly-L-lactic acid. J Cosmet Dermatol Sci Appl 2012;2:20
- [Background] Orringer JS, Kang S, Johnson TM, Karimipour DJ, Hamilton T, Hammerberg C, Voorhees JJ, Fisher GJ. Connective tissue remodeling induced by carbon dioxide laser resurfacing of photodamaged human skin. Arch Dermatol. 2004 Nov;140(11):1326-32. doi: 10.1001/archderm.140.11.1326. PMID 15545540
- [Background] Branham GH, Thomas JR. Rejuvenation of the skin surface: chemical peel and dermabrasion. Facial Plast Surg. 1996 Apr;12(2):125-33. doi: 10.1055/s-0028-1082404. PMID 9220727
- [Background] Nikolis A, Bernstein S, Kinney B, Scuderi N, Rastogi S, Sampalis JS. A randomized, placebo-controlled, single-blinded, split-faced clinical trial evaluating the efficacy and safety of KLOX-001 gel formulation with KLOX light-emitting diode light on facial rejuvenation. Clin Cosmet Investig Dermatol. 2016 May 13;9:115-25. doi: 10.2147/CCID.S100697. eCollection 2016. PMID 27257391
- [Background] Airan LE, Hruza G. Current lasers in skin resurfacing. Facial Plast Surg Clin North Am. 2005 Feb;13(1):127-39. doi: 10.1016/j.fsc.2004.06.005. PMID 15519933